CLINICAL TRIAL: NCT05751759
Title: A Phase I Single Dose, Non-Randomised, Open-Label, Parallel Group Study to Investigate the Effect of Hepatic Impairment on the Pharmacokinetics, Safety and Tolerability of Mitiperstat
Brief Title: Pharmacokinetics of Mitiperstat in Participants With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6581C00002
Record Dates: First submitted 2023-02-21; First posted 2023-03-02 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Hepatic Impairment
Keywords: Hepatic impairment; Liver disease
MeSH Terms: conditions — Liver Diseases | interventions — AZD4831

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): 8 participants with mild hepatic impairment (Child-Pugh A) will be given Dose A of mitiperstat.
  Interventions: Drug: Mitiperstat
- Cohort 2 (Experimental): 8 participants with moderate hepatic impairment (Child-Pugh B) will be given Dose A of mitiperstat.
  Interventions: Drug: Mitiperstat
- Cohort 3 (Experimental): 6-8 participants with severe hepatic impairment (Child-Pugh C) will be given Dose A of mitiperstat.
  Interventions: Drug: Mitiperstat
- Cohort 4 (Experimental): 8-12 participants with normal hepatic function will be given Dose A of mitiperstat.
  Interventions: Drug: Mitiperstat

INTERVENTIONS:
Drug: Mitiperstat — Participants receive mitiperstat orally.
  Other Names: AZD4831

SUMMARY:
This study will assess the effect of hepatic impairment on the pharmacokinetics (PK), safety and tolerability of mitiperstat.

DETAILED DESCRIPTION:
This is a Phase I, single dose, non-randomised, open-label, parallel group study to examine the PK, safety, and tolerability of mitiperstat in participants with hepatic impairment and participants with normal hepatic function.

Participants will be assigned to one of the following cohorts as per Child-Pugh classification:

* Cohort 1: Eight participants with Mild hepatic impairment (Child-Pugh A)
* Cohort 2: Eight participants with Moderate hepatic impairment (Child-Pugh B)
* Cohort 3: Six to eight participants with Severe hepatic impairment (Child-Pugh C)
* Cohort 4: Eight to twelve participants with Normal hepatic function

A final safety follow-up visit on Day 21 will be there after all procedures are completed on Day 15.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥ 18 to ≤ 85 years (inclusive), at the time of signing the informed consent.
* Weight ≥ 50kg and BMI ≥ 18 kg/m2 up to < 42 kg/m2.
* Male and/or females.
* Contraceptive use by females should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

  1. Criterion not applicable to this CSP version.
  2. Female participants:

     * Female participants must not be lactating.
     * Female participants of childbearing potential who are sexually active with a non-sterilised male partner must agree to use an acceptable method of birth control, from enrolment throughout the study and until at least 4 weeks after the last dose of study intervention.
* Capable of giving signed informed consent.

Participants with hepatic impairment only:

* Supporting documents confirming that the participant has liver cirrhosis with hepatic impairment must be available.
* Diagnosis of chronic and stable hepatic impairment.

Exclusion Criteria:

* Any positive result on screening for serum or plasma hepatitis B surface antigen, hepatitis C antibody, and HIV.
* History of substance dependence or a positive screen for drugs of abuse, likely to impact participant safety or compliance with study procedures.
* History of alcohol abuse or excessive intake of alcohol in the last 12 months.
* Abnormal vital signs, after 10 minutes supine rest at screening or Day -1.
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting 12-lead ECG at screening or Day -1:
* Vulnerable participants.
* For female participants only: currently pregnant or breast-feeding.

Participants with hepatic impairment only

* Participants with previous transjugular intrahepatic portosystemic shunt (TIPS).
* Severe ascites defined as ascites requiring paracentesis and albumin at 4-week intervals or less.
* Fluctuating or rapidly deteriorating hepatic function, as indicated by strongly varying or worsening of clinical and/or laboratory signs of hepatic impairment within the screening period.
* Any evidence of additional severe or uncontrolled systemic disease or laboratory finding that makes it unsafe for the participant to participate in the study.
* Change in dose regimen of medically-required medication within the last 2 weeks before pre-study examination.
* Biliary obstruction or other causes of hepatic impairment not related to parenchymal disorder and/or disease of the liver.
* Clinically relevant hepatic encephalopathy.
* Oesophageal variceal bleeding in prior 3 months.
* Platelet count < 50 × 109/L and/or neutrophil count < 1.2 × 109/L and/or haemoglobin < 85 g/L.
* Post liver transplantation.
* History of acute or chronic pancreatitis, or pancreatic amylase or lipase greater than twice the ULN at screening.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2024-11-21 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Day 1 to Day 15
  The Cmax of a single dose of mitiperstat in participants with impaired hepatic function and controls with normal hepatic function will be evaluated and compared.
Area under the concentration-time curve from time zero to infinity (AUCinf) | Day 1 to Day 15
  The AUCinf of a single dose of mitiperstat in participants with impaired hepatic function and controls with normal hepatic function will be evaluated and compared.
Area under the concentration-time curve from time zero to last time of quantifiable concentration (AUClast) | Day 1 to Day 15
  The AUClast of a single dose of mitiperstat in participants with impaired hepatic function and controls with normal hepatic function will be evaluated and compared.
Apparent terminal elimination half-life (t½λz) | Day 1 to Day 15
  The t½λz of a single dose of mitiperstat in participants with impaired hepatic function and controls with normal hepatic function will be evaluated.
Time to Cmax (tmax) | Day 1 to Day 15
  The tmax of a single dose of mitiperstat in participants with impaired hepatic function and controls with normal hepatic function will be evaluated.
Apparent Clearance (CL/F) | Day 1 to Day 15
  The CL/F of a single dose of mitiperstat in participants with impaired hepatic function and controls with normal hepatic function will be evaluated.
Volume of distribution (apparent) following extravascular administration [based on terminal phase] (Vz/F) | Day 1 to Day 15
  The Vz/F of a single dose of mitiperstat in participants with impaired hepatic function and controls with normal hepatic function will be evaluated.
Cumulative amount of unchanged drug excreted into urine (Ae[0-24]) | Day 1 to Day 15
  The Ae(0-24) of a single dose of mitiperstat in participants with impaired hepatic function and controls with normal hepatic function will be evaluated.
Renal clearance of drug from plasma (CLR) | Day 1 to Day 15
  The CLR of a single dose of mitiperstat in participants with impaired hepatic function and controls with normal hepatic function will be evaluated.
Non-renal clearance of drug from plasma (CLNR) | Day 1 to Day 15
  The CLNR of a single dose of mitiperstat in participants with impaired hepatic function and controls with normal hepatic function will be evaluated.
Percentage of dose excreted unchanged in urine from time 0 to time 24 (fe[0-24) | Day 1 to Day 15
  The fe(0-24) of a single dose of mitiperstat in participants with impaired hepatic function and controls with normal hepatic function will be evaluated.

SECONDARY OUTCOMES:
Adverse Events (AEs), and Serious Adverse Events (SAEs) | From time of dose to the final follow-up visit (Day 21 [± 4 days])
  The safety, and tolerability of a single dose of mitiperstat in participants with hepatic impairment and controls with normal hepatic function will be assessed.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Research Site, Rialto, California
  - Research Site, Hialeah, Florida
  - Research Site, Orlando, Florida
  - Research Site, Canton, Ohio
  - Research Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual participant-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home